CLINICAL TRIAL: NCT00734175
Title: Phase I Inpatient Study of the Safety and Immunogenicity of Live Influenza A Vaccine H6N1 (6-2) AA ca Recombinant (A/Teal/Hong Kong/W312/1997 (H6N1) x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Avian Influenza H6N1 Infection in the Event of a Pandemic
Brief Title: Safety of and Immune Response to Recombinant Live-Attenuated Influenza H6N1 Virus Vaccine Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Kawsar Talaat, MD, Johns Hopkins Bloomberg School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 251
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2008-09

CONDITIONS: Influenza; Virus Diseases
Keywords: Vaccine; Influenza
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participants will receive 2 doses of vaccine 4 to 8 weeks (28-62 days) apart
  Interventions: Biological: H6N1 Teal HK 97/AA ca recombinant vaccine

INTERVENTIONS:
Biological: H6N1 Teal HK 97/AA ca recombinant vaccine — Approximately 0.2 ml of 10^7 TCID50 doses of vaccine administered intranasally

SUMMARY:
In the 20th century, influenza pandemics occurred in 1918, 1957, and 1968, and were associated with significant morbidity and mortality. It is estimated that, in the United States alone, the next influenza pandemic could cause approximately 200,000 deaths and 750,000 hospitalizations. Thus, the development of a vaccine against potential influenza strains has become a priority. The purpose of this study is to determine the safety and immune response to an H6N1 influenza vaccine candidate.

DETAILED DESCRIPTION:
H6 influenza viruses are of the low pathogenicity phenotype in poultry, and in the last decade, outbreaks of H6 influenza infection have been reported both in the United States and South Africa. The prevalence of H6 influenza viruses in a wide range of domestic and wild birds, and their propensity for reassortment has raised concerns regarding the pandemic potential of these viruses. This vaccine, therefore, is an important priority in the development of vaccines against potential pandemic influenza strains.

This vaccine trial will be conducted in the Center for Immunization Research inpatient unit in the Mason F. Lord Building at the Johns Hopkins Bayview Medical Center (Baltimore, MD). The study will be initiated between April 1st and December 20th, 2008, when wild-type influenza is unlikely to be circulating in the Baltimore area.

An individual's participation in the study will last approximately 90 days. All participants will receive two vaccinations approximately 4 - 8 weeks apart. After each vaccination, participants will remain in isolation at the study site for at least nine days or until rRT-PCR assays for influenza are negative for 2 consecutive days. A physical examination and nasal wash will occur each day during the isolation period. Blood collection will occur on the day of admission, the following day, and day 7 after vaccination. Follow-up outpatient visits are scheduled on Days 28 and 56 after the first vaccination and on Day 28 after the second vaccination. Follow-up visits will include serum collection, nasal wash, and interim medical history.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females 18-49 years old
* General good health
* Available for the duration of the trial
* If female, agree to use effective birth control methods for the duration of the study. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease. More information on this criterion can be found in the protocol.
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, intereferes with the study
* Previous receipt of FluMist or any intranasal live attenuated influenza vaccine
* Previous enrollment in an H6N1 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H6N1 influenza A virus (serum HAI titer >1:8)
* Positive urine drug toxicology test indicating narcotic use and/or dependency as defined by the Drug Enforcement Agency
* Medical, occupational, or family problems as a result of alcohol or illicit drug use within the 12 months prior to study entry
* Any condition that, in the opinion of the investigator, would interfere with the study
* History of anaphylaxis
* Allergy to oseltamivir as determined by subject report
* Current diagnosis of asthma or reactive airway disease within 2 years prior to study entry
* History of Guillain-Barre Syndrome
* HIV-1-infected
* Hepatitis C-infected
* Positive hepatitis B virus surface antigen
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to study entry
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study entry
* History of a surgical splenectomy
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study entry
* Current smoker unwilling to stop smoking for the duration of the study. More information on this criterion can be found in the protocol.
* Travel to the Southern Hemisphere within 14 days prior to study entry
* Travel on a cruise ship within 14 days prior to study entry
* Direct contact with live poultry within the 14 days prior to the study or after study completion.
* Receipt of another investigational vaccine or drug within 30 days prior to study entry
* Allergy to eggs or egg products
* Pregnant or breastfeeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events and other adverse events | Throughout study
Amount of vaccine virus shed by each participant | Throughout study
Amount of serum and nasal wash antibody induced by the vaccine | Throughout study

SECONDARY OUTCOMES:
Number of participants infected with the H6N1 Teal HK 97/AA ca recombinant vaccine | Throughout study
Phenotypic stability of vaccine virus shed | Throughout study
Determine whether immunogenicity is enhanced by a second dose of vaccine, and whether the first dose of vaccine restricts replication of the second dose | Throughout study
T-cell mediated and innate immune responses against the H6N1 Teal HK 97/AA ca recombinant vaccine | Throughout study
Development of serum bank so that the capacity of the H6N1 Teal HK 97/AA ca recombinant vaccine to elicit HA1 and neutralizing antibodies to future H6 influenza viruses can be tested | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bayview Medical Center, CIR Unit at the Mason F Lord Building, Baltimore, Maryland, United States

REFERENCES:
- [Background] Eichelberger M, Golding H, Hess M, Weir J, Subbarao K, Luke CJ, Friede M, Wood D. FDA/NIH/WHO public workshop on immune correlates of protection against influenza A viruses in support of pandemic vaccine development, Bethesda, Maryland, US, December 10-11, 2007. Vaccine. 2008 Aug 12;26(34):4299-303. doi: 10.1016/j.vaccine.2008.06.012. Epub 2008 Jun 26. PMID 18582523
- [Background] Hampson AW. Vaccines for pandemic influenza. The history of our current vaccines, their limitations and the requirements to deal with a pandemic threat. Ann Acad Med Singap. 2008 Jun;37(6):510-7. PMID 18618064
- [Background] Wright PF. Vaccine preparedness--are we ready for the next influenza pandemic? N Engl J Med. 2008 Jun 12;358(24):2540-3. doi: 10.1056/NEJMp0803650. No abstract available. PMID 18550873
- [Derived] Talaat KR, Karron RA, Luke CJ, Thumar B, McMahon BA, Chen GL, Lamirande EW, Jin H, Coelingh KL, Kemble G, Subbarao K. An open label Phase I trial of a live attenuated H6N1 influenza virus vaccine in healthy adults. Vaccine. 2011 Apr 12;29(17):3144-8. doi: 10.1016/j.vaccine.2011.02.043. Epub 2011 Mar 4. PMID 21377509